CLINICAL TRIAL: NCT00737204
Title: Armodafinil Treatment for Fatigue in HIV+ Patients
Brief Title: Effectiveness of Armodafinil for Treating Fatigue in Adults With HIV/AIDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #4839/5892R; R01MH072383-02 (NIH)
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2013-03

CONDITIONS: HIV Infections; Fatigue
Keywords: HIV; AIDS; Armodafinil; Depression
MeSH Terms: conditions — HIV Infections; Fatigue; Acquired Immunodeficiency Syndrome; Depression | interventions — Modafinil; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Armodafinil (Experimental): Participants will take armodafinil for 4 weeks. The dose will be titrated up from 50mg to 250mg per day as clinically indicated, using 50mg tablets. If responsive, participants will be offered 12 additional weeks of armodafinil.
  Interventions: Drug: Armodafinil
- Placebo (Placebo Comparator): Participants will receive placebo pills for 4 weeks. Placebo tablets that match the 50mg active medication tablets will given following the same dosing strategy as Arm 1. The dose will be titrated from 1 placebo tablet daily to 5 tablets daily as clinically indicated. Non-responders to placebo will then be offered 16 weeks of active medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Armodafinil — Participants will receive 50 mg of armodafinil per day, increasing to 250 mg per day as clinically indicated.
  Other Names: Nuvigil
  Arms: Armodafinil
Drug: Placebo — Participants will receive placebo pills matched to the active armodafinil and according to the same dosing strategy
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This study will determine whether armodafinil (Nuvigil), an FDA approved medication, is effective in reducing fatigue in adults with HIV/AIDS.

DETAILED DESCRIPTION:
Fatigue is a common problem for many people with HIV/AIDS, interfering with daily activities and serving as a significant barrier to working among those whose health is otherwise stable or restored by antiretroviral (ARV) medication. Fatigue in HIV is associated with disability and diminished quality of life. It may be caused by ARVs or by the virus itself. A related study tested whether modafinil, of which armodafinil is an r-isomer, could reduce fatigue in HIV/AIDS patients. Armodafinil, believed to have a longer duration and greater effect than modafinil, will be tested on the same criteria.

Participants will be randomly assigned to receive either armodafinil or a placebo daily for 4 weeks. Participants randomized to active medication and who show improvements in symptoms will be offered armodafinil for an additional 12 weeks. For them, the study duration is 16 weeks. Participants who did not receive armodafinil will be offered armodafinil for 16 weeks. For these participants, the study duration is 20 weeks. Participants who did not benefit from armodafinil will receive alternate treatment options. All participants will have weekly study visits for the first 4 weeks of the study and biweekly visits for the remainder of the study. At each visit, participants will complete various tasks to determine cognitive function, and self-report scales will be used to determine symptoms of depression and fatigue. After completion of 16 weeks, participants responding to armodafinil will be transitioned to the publicly available modafinil over the course of 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-75
2. HIV+
3. Clinically significant fatigue (score of 4.5+ on Fatigue Severity Scale, plus impairment on 1+ categories of Role Function Scale)
4. Fatigue duration for 3+ months
5. English-speaking
6. Able to give informed consent
7. Fecund women uses barrier method of contraception

Exclusion Criteria:

1. Primary care doctor does not approve of study participation
2. Unstable medical condition (e.g. liver failure; cirrhosis, new onset opportunistic infection in past month)
3. Untreated hypogonadism, except for men for whom testosterone replacement is medically contraindicated (serum testosterone below the reference range)
4. Untreated hypothyroidism (Thyroid Stimulating Hormone over 5 IUI/mL)
5. Untreated and uncontrolled hypertension
6. Clinically significant anemia (hematocrit <30%)
7. Started testosterone or nandrolone in past 6 weeks
8. Started or changed an antiretroviral regimen in past 4 weeks if fatigue predated the change; otherwise, started or changed regimen in past 2 months
9. Untreated or under-treated major depressive disorder
10. Started antidepressant medication within past 6 weeks
11. Substance abuse/dependence (past 4 months)
12. Regular and frequent cannabis use (> twice/week regularly)
13. Currently clinically significant suicidal ideation or Hamilton Depression Scale (HAM-D) score >24
14. History or current psychosis or bipolar disorder
15. Pregnant or breastfeeding
16. Significant untreated insomnia (score >3 on HAM-D insomnia items)
17. Currently taking psychostimulant medication or past nonresponse to modafinil
18. Has no alternative viable antiretroviral regimen after the current one
19. Left ventricular hypertrophy; mitral valve prolapse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-06; Primary Completion 2010-04 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith G. Rabkin, Phd, MPH, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Background] Rabkin JG, McElhiney MC, Rabkin R, Ferrando SJ. Modafinil treatment for fatigue in HIV+ patients: a pilot study. J Clin Psychiatry. 2004 Dec;65(12):1688-95. doi: 10.4088/jcp.v65n1215. PMID 15641875
- [Result] Rabkin JG, McElhiney MC, Rabkin R. Treatment of HIV-related fatigue with armodafinil: a placebo-controlled randomized trial. Psychosomatics. 2011 Jul-Aug;52(4):328-36. doi: 10.1016/j.psym.2011.02.005. PMID 21777715

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from community based organizations and healthcare clinics that provide services to persons with HIV, by placing flyers on bulletin boards and in waiting areas.
Pre-assignment Details: A total of 114 patients were screened for eligibility, 25 had medical or psychiatric exclusion criteria, 7 were active substance users, 4 were taking stimulants, 3 were not clinically fatigued, 5 declined participation, and 70 were randomized. Of the 70, 64 completed the 4-week trial.
Groups:
- Armodafinil: Participants will receive armodafinil for 4 weeks. If responsive, participants will be offered 12 additional weeks of armodafinil. Starting dose of armodafinil is 50 mg/day, increased weekly in the absence of clinical response and dose-limiting side effects to a maximum of 250 mg/day.
- Placebo: Participants will receive a placebo pill (matching the active medication) for 4 weeks, then a 16-week course of armodafinil. Starting dose of is one placebo pill/day, increased weekly in the absence of clinical response and dose-limiting side effects to a maximum of 5 placebo pills/day.
Period: Overall Study
Arm/Group | Armodafinil | Placebo
Started | 36 | 34
Completed | 36 | 28
Not Completed | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Armodafinil: Participants will receive armodafinil for 4 weeks. If responsive, participants will be offered 12 additional weeks of armodafinil.
- Placebo: Participants will receive a placebo pill for 4 weeks, then a 16-week course of armodafinil.
- Total: Total of all reporting groups
Arm/Group | Armodafinil | Placebo | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 34 | 70
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (8.7) | 46 (8.2) | 46 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 31 | 30 | 61
Region of Enrollment [Number; unit: participants]
  United States | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Severity Scale(FSS) Outcome
Description: The FSS is a 9-item self-report scale that measures the impact of fatigue on everyday functioning. Each item is rated on a scale of 1 to 7. Total scores range from 9-63, with a higher score indicating greater impairment due to fatigue.
Time Frame: Measured at baseline and Weeks 4
Population: Of the 70 patients randomized, 64 completed the 4-week trial. Data presented are for the 70, using the last data point carried forward (intention to treat).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 36 | 34
units on a scale
  Baseline FSS | 52.6 (6.13) | 53.1 (6.87)
  Week 4 FSS | 25.8 (14.23) | 39.4 (14.91)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Primary Outcome: Role Function Scale
Description: The Role Function Scale includes 10 items drawn from the Short Form 36-item Survey (SF-36) and other SF versions. It is intended to assess the extent to which fatigue has a behavioral impact on daily activities. Scores of frequency in the past week, on a 5-point scale, are summed with higher scores signifying greater role impairment. Scores range from 10-50.
Time Frame: Measured at Baseline and Week 4
Population: The week 4 outcome analyses are based on an intention to treat sample, which includes the 6 dropouts, using the last data point brought forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 36 | 34
units on a scale
  Baseline Role Function Scale | 36.2 (5.75) | 37.8 (7.81)
  Week 4 Role Function Scale | 19.9 (8.1) | 28.3 (10.19)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Repeated measure analysis; Test type: Superiority or Other; p = .01, ANCOVA

3. Secondary Outcome: CD4 Cell Count
Description: Cd4 cell count is a laboratory marker providing an indication of immune system functioning. Blood samples were drawn for this measure at baseline and week 4. The reference range for CD4 cell count is 490-1740, and a clinically significant change is defined as a change of >=100 cells. A higher number is associated with better immune functioning.
Time Frame: Measured at baseline and Week 4
Population: Results were included for patients on whom baseline and week 4 labs were drawn.
Measure: Mean (Standard Deviation); unit: Cells/mcL
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 35 | 27
Cells/mcL
  Baseline CD4 cell count | 502 (202) | 450 (241)
  Week 4 CD4 cell count | 503 (224) | 445 (255)
Statistical Analysis 1: Comparison: Armodafinil vs Placebo; Null hypothesis: CD4 levels for both the Armodafinil and Placebo groups will not change significantly between baseline and week 4; Test type: Superiority or Other; p >= .805, Paired t-tests

4. Secondary Outcome: HIV Viral Load
Description: HIV RNA viral load assay is a laboratory measure indicating viral activity. Because of the large range of possible values (50 - 100,000 copies), this measure is transformed to log10 values. We entered the log10 value of 1.69 when the laboratory result stated "under 50 copies," which was the assay's lowest limit of detectability during the study.
Time Frame: Measured at baseline and Week 4
Population: Results were included for patients on whom baseline and week 4 labs were drawn.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | Armodafinil | Placebo
Number analyzed (Participants) | 36 | 27
Log10 copies/mL
  Baseline Log10 Viral Load | 2.17 (0.81) | 2.39 (1.13)
  Week 4 Log10 Viral load | 2.15 (0.87) | 2.24 (1.07)

ADVERSE EVENTS:
Time Frame: Treatment emergent side effects were assessed at baseline and then weekly during the 4-week trial.
Description: Each potential side effect was rated on a 0 ("No Problems" to 5 ("Severe Problems"). An increase of 2 points during the trial from the baseline score was considered an adverse event.
Arm/Group | Armodafinil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 0/36 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No